CLINICAL TRIAL: NCT06774716
Title: Internet-delivered Cognitive Behavior Therapy for Problematic Alcohol Use in a Working Life Setting: a Research Protocol for Qualitative and Quantitative Evaluation of Feasibility and Outcomes
Brief Title: Internet-delivered Cognitive Behavior Therapy for Problematic Alcohol Use in a Working Life Setting
Acronym: Simba
Status: Completed | Type: Observational
Sponsor: Stockholm University (Other)
Collaborators: AFA Insurance (Industry); Systembolagets alkoholforskningsråd (Unknown); Alna Sverige AB (Unknown); Karolinska Institutet (Other); Uppsala University (Other)
Responsible Party: Principal Investigator, Kristina Sundqvist, PhD, Stockholm University
Other Study IDs: 1800008
Record Dates: First submitted 2022-05-10; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Use Disorder; Alcohol Abuse
Keywords: Problematic alcohol use; Work life; Cognitive Behavior Therapy; Feasibility; Outcome; Employee assistance program; Internet; qualitative; quantitative
MeSH Terms: conditions — Alcoholism | interventions — Secondary Prevention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ICBT: Internet-based cognitive behaviour treatment, based on relapse prevention, delivered in a work-life setting.
  Interventions: Behavioral: Internet-based cognitive behavioural treatment and relapse prevention
- Face-to-face treatment as ususal: Face-to-face treatment as usual, based on relapse prevention, delivered in a work-life setting.
  Interventions: Behavioral: Face-to-face cognitive behavioural treatment or short-term psycodynamic therapy with relapse prevention

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioural treatment and relapse prevention — A self help program consisting of 12 modules and access to therapist guidance through messages. Including three video session.
  Groups: ICBT
Behavioral: Face-to-face cognitive behavioural treatment or short-term psycodynamic therapy with relapse prevention — Face-to-face therapy with a licenced psychologist or licenced psychotherapist, including 10-15 sessions.
  Groups: Face-to-face treatment as ususal

SUMMARY:
Internet-based cognitive behavioral treatment (ICBT) for mental health issues has been successfully implemented in routine health care and research indicates that ICBT can also be applied to decrease problematic alcohol use in healthcare as well as working life settings. However, qualitative studies investigating the feasibility of implementing ICBT in a working life context have been lacking. The current study will investigate the feasibility of delivering ICBT for problematic alcohol use within an employee assistance program (EAP), and will compare outcomes for ICBT with face-to-face treatment in a naturalistic quantitative study. Recruitment to the study follows employer contact with the EAP regarding an employee's presumed problematic alcohol consumption, leading to a five-session in-person psychological assessment. All assessed employees recommended ICBT or face-to-face treatment will be offered participation in the study. In addition to quantitative evaluation, interviews will be conducted with employees and their employer representatives following ICBT to elucidate both stakeholders' experience and perception of ICBT in the work life context. Thematic analysis and grounded theory will be used to analyze the interview material. Outcome comparisons between ICBT and face-to-face treatment will be assessed quantitatively using a Reliable Change Index and analysis of variance or other relevant statistical analyses such as multilevel modeling.

ELIGIBILITY:
Inclusion Criteria:

18 years; access to the Internet; problematic alcohol use assessed by a licenced psychologist; referred to treatment within a rehabilitation intervention initiated by the work-place; Work-place covers treatment costs;

Exclusion Criteria:

not adequately fluent in Swedish; drug use; suicidality; indications of excessive use of the internet and computer gaming and/or gambling;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Employees that have undergone an assessment as a rehabilitation intervention initiated by the employer. Participants included have a problematic alcohol use, and are referred to treatment where the employer covers the cost of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back (TLFB) | Baseline and 14 weeks, 6 months, 12 months and
  Change in total TLFB score (consumption during preceding week), as a summarized measure of alcohol consumption

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | Baseline and 14 weeks, 6 months, 12 months
  Change in total AUDIT score, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems)
Patient Health Questionnaire (PHQ-9) | Baseline and 14 weeks, 6 months, 12 months
  Change in total PHQ-9 score, as a summarized measure of depression
Generalized Anxiety Disorder-7 (GAD-7) | Baseline and 14 weeks, 6 months, 12 months
  Change in total GAD-7 score, as a summarized measure of anxiety
The WHO-5 well-being-index | Baseline and 14 weeks, 6 months, 12 months
  Change in total WHO-5 score, as a summarized measure of general well-being

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Sundqvist, PhD, Principal Investigator — Stockholm University
Locations (1):
- Stockholm University, Stockholm, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: No